CLINICAL TRIAL: NCT04842370
Title: A Prospective, Phase Ia/Ib, Multicenter Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of the FLT3 Inhibitor, PHI 101, Alone in Subjects With Relapsed or Refractory Acute Myeloid Leukemia (AML)
Brief Title: Evaluation of the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of PHI 101 for the Treatment of AML
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Collaborators: Pharos iBio Co., Ltd. (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PHI-101-001
Record Dates: First submitted 2021-04-08; First posted 2021-04-13 (Actual); Last update posted 2021-04-20 (Actual); Status verified 2021-04

CONDITIONS: Relapsed or Refractory Acute Myeloid Leukemia
MeSH Terms: conditions — Recurrence; Leukemia, Myeloid, Acute | interventions — PHI-101

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dose escalation and expansion of PHI-101 (Experimental)
  Interventions: Drug: PHI-101

INTERVENTIONS:
Drug: PHI-101 — PHI-101, oral, once-daily administration, consisting of 28-days per 1 cycle

SUMMARY:
The purpose of this study is to find out the maximum tolerable dose and safety of PHI-101, novel FLT3 inhibitor in the treatment of relapsed or refractory AML for patients who have received standard therapy or cannot tolerate standard therapy, and/or for whom no standard therapy exists.

There will be two parts to the study, which we will call Phase Ia and Phase Ib. Phase Ia is called the dose escalation. Approximately 20 to 24 patients are planned to be enrolled into Phase Ia. Phase 1a is conducted to determine the best dose and schedule of dosing of PHI-101 to be used in Phase 1b. There will be 5 different dose levels of PHI-101 given to patients in Phase Ia.

Phase Ib is called the dose expansion. Approximately 14-34 patients (approximately 14-17 patients in each of the 2 cohorts planned) of each cohort are planned in Phase Ib based on study design. Phase Ib is also being conducted to assess anti-leukemia response, changes in transfusion requirements, and safety of PHI-101 at the dose level identified during Phase Ia.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to understand and sign an informed consent form (ICF) and to comply with all aspects of the protocol.
* Female or male subjects aged ≥18 years of age.
* The ECOG performance status ≤2.
* Life expectancy more than 3 months.
* Phase Ia (dose escalation part only): Subjects with relapsed and/or refractory AML which is diagnosed with World Health Organization (WHO) classification9 who have received standard therapy or are intolerant of standard therapy, and/or for whom no standard therapy exists.
* Phase Ib (dose expansion): Subjects with relapsed and/or refractory AML which is diagnosed with WHO classification and who have a FLT3 abnormality (i.e., FLT3-ITD and/or TKD mutation) as determined by accredited laboratory.
* Female subjects must be surgically sterile, or have a monogamous partner who is surgically sterile, or be of postmenopausal status (at least 2 years or serum follicle stimulating hormone >40 mIU/mL and estradiol <20 pg/mL or according to the postmenopausal range definition for the laboratory involved), or commit to use an effective form of birth control (Appendix 5) for the duration of the study and for 90 days following the last PHI-101 administration.
* Sexually active males must commit to use an effective form of birth control (Appendix 5) while taking the drug and for 30 days after stopping PHI-101. A condom is required to be used by vasectomized men in order to prevent delivery of the drug via seminal fluid.
* Subject having laboratory values defined as:

Creatinine clearance (calculated using Cockcroft-Gault formula, or measured) >40 mL/min.

Total bilirubin <1.5 × upper limit of normal (ULN), except for subjects with Gilbert's syndrome who are excluded if total bilirubin >3.0 × ULN or direct bilirubin ≥1.5 × ULN.

Alanine aminotransferase (ALT) <2.5 × ULN, except for subjects that have leukemic involvement of the liver, who are excluded if ALT <5 × ULN.

Aspartate aminotransferase (AST) <2.5 × ULN, except for subjects that have leukemic involvement of the liver, who are excluded if AST <5 × ULN.

Exclusion Criteria:

* Presence of overt leptomeningeal or active central nervous system involvement with AML.
* Subject has a diagnosis of acute promyelocytic leukemia (APL), French American British classification M3 or WHO classification of APL with t(15;17)(q22;q12), or BCR ABL positive leukemia (chronic myelogenous leukemia in blast crisis).
* Subject has favorable risk cytogenetics as categorized by the National Comprehensive Cancer Network Guidelines Version 2, 2014 for AML.
* Subject has had hematopoietic stem cell transplant and meets any of the following:

Is within 2 months of transplant from Cycle 1 Day 1. Has clinically significant Graft-versus-host disease requiring treatment. Has ≥ Grade 2 persistent nonhematological toxicity related to the transplant. Donor lymphocytes infusion is not permitted ≤30 days prior to study registration or during the first cycle of treatment.

* Subject has disseminated intravascular coagulation abnormality.
* Impaired cardiac function or clinically significant cardiac disease, including any of the following:

Clinically significant and/or uncontrolled heart disease such as congestive heart failure requiring treatment (New York Heart Association Grade ≥2), left ventricular ejection fraction <50% as determined by multiple gated acquisition (MUGA) or echocardiogram, uncontrolled hypertension, or clinically significant arrhythmia.

QT interval as corrected by the Fridericia method (QTcF) >450 ms ECG or congenital long QT syndrome at the Screening Visit.

Subject with hypokalemia and hypomagnesemia at Screening (defined as values below lower limit of normal).

Acute myocardial infarction or unstable angina pectoris <3 months prior to study entry.

* Subjects with interstitial pneumonia or history of drug-induced interstitial pneumonia/pneumonitis.
* A positive human immunodeficiency virus (HIV) antibody test.
* Active hepatitis B virus (HBV) infection (chronic or acute), defined as having a positive hepatitis B surface antigen (HBsAg) test, or active hepatitis C virus (HCV) infection, defined as having a positive HCV antibody test followed by a positive HCV RNA test.

Note: Subjects with a past or resolved HBV infection, defined as having a negative HBsAg test and a positive hepatitis B core antibody test followed by a quantitative HBV DNA < 9 log (80) IU/mL are eligible for the study. Subjects who are inactive carriers of HBV/HCV are eligible for the study.

* Chronic liver disease or chronic hepatitis (Child Pugh Class B or C hepatic impairment).
* Any gastrointestinal disorders interfering with study drug absorption or subjects who are unable to swallow tablets or capsules.
* Malignant disease, other than that being treated in this study. Exceptions to this exclusion include the following: malignancies that were treated curatively and have not recurred within 2 years prior to study treatment; completely resected basal cell and squamous cell skin cancers; any malignancy considered to be indolent and that has never required therapy; and completely resected carcinoma in situ of any type.
* Subjects receiving systemic chronic steroid therapy or any immunosuppressive therapy (≥10 mg/day prednisone or equivalent). Topical, inhaled, nasal, and ophthalmic steroids are allowed.
* Use of any live vaccines against infectious diseases within 28 days of initiation of study treatment.
* Use of medications, herbal products, or foods known to be moderate or potent inhibitors of P glycoprotein (P gp) within the last 7 days prior to Day 1 or known to be moderate or potent inducers of P gp within the last 14 days prior to Day 1 (see Section 6.5).
* Subjects with a history of stroke or having active neurological symptoms, with the exception of chronic conditions which in the opinion of the neurologist, Investigator, and the Sponsor, would not impact on ongoing neurologic assessments while on study treatment.
* Active uncontrolled infection requiring systemic or antiviral antibiotic therapy.
* Major surgery within 2 weeks of the first dose of study treatment (mediastinoscopy, insertion of a central venous access device, and insertion of a feeding tube are not considered major surgery).
* Radiotherapy within 3 weeks of the first dose of study drug, except for palliative radiotherapy to a limited-field, such as for the treatment of bone pain or a focally painful tumor mass.
* Presence of CTCAE ≥ Grade 2 toxicity (except alopecia, peripheral neuropathy, and ototoxicity, which are excluded if ≥ CTCAE Grade 3) due to prior cancer therapy.
* Prior treatment with cytotoxic agents (except hydroxyurea given for controlling hyperleukocytosis) within 2 weeks prior to study drug administration, or other experimental agents or noncytotoxic agents within 5 half-lives prior to study drug administration.

Note: Subjects in Phase Ia of this study can still take PHI-101 before entering Phase Ib of this study.

* Any medical condition that would, in the Investigator's judgment, prevent the subject's participation in the clinical study due to safety concerns, compliance with clinical study procedures, or interpretation of study results.
* Pregnant or lactating women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive human chorionic gonadotropin laboratory test.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2020-06-08 (Actual); Primary Completion 2022-05-21 (Estimated); Study Completion 2022-05-21 (Estimated)

PRIMARY OUTCOMES:
Safety assessed through adverse events to determine maximum tolerated dose | From screening to the last Safety Follow up Visit(Safety Follow-up visit occurs 30 days after from EOT)
  Safety will be measured by AEs, vital signs, ECG, clinical laboratory tests, physical examination, ECOG performance.
Tolerability assessed by dose compliance | From screening to the last Safety Follow up Visit(Safety Follow-up visit occurs 30 days after from EOT)
  Tolerability will be measured by reviewing data of dose interruptions, reductions, and doses administered

CONTACTS AND LOCATIONS:
Overall Officials: Sung-Soo Yoon, MD. PhD, Principal Investigator — Seoul National University Hospital, Seoul National University College of Medicine
Locations (1):
- Seoul National University Cancer Hospital, Seoul, South Korea